CLINICAL TRIAL: NCT07387029
Title: Core Stability Training With Ball and Balloon Exercise on Dynamic Balance, Hop Performance, and Core Endurance in Professional Football Players - A Randomized Clinical Trial
Brief Title: Core Stability Training With Balloon Breathing on Balance and Performance in Football Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-COHS-STD-117-Dec-2025
Record Dates: First submitted 2026-01-22; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Dynamic Balance, Hop Performance and Maximum Voluntary Ventilation (MVV) in Professional Football Players
Keywords: Dynamic balance; Diaphragmatic breathing; Core stability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stability Training With Balloon Breathing (Experimental): Participants receive a structured core stability training program combined with balloon breathing exercises along with regular football training for 8 weeks.
  Interventions: Other: Core Stability Training; Other: Balloon Breathing Exercise
- Core Stability Training Only (Active Comparator): Participants receive the same structured core stability training program without balloon breathing exercises, along with regular football training for 8 weeks.
  Interventions: Other: Core Stability Training

INTERVENTIONS:
Other: Core Stability Training — McGill's Big Three core stability exercises including curl-up, side bridge, and bird-dog exercises performed three times per week for eight weeks, with progression to unstable surfaces as tolerated.
Other: Balloon Breathing Exercise — Diaphragmatic breathing exercise involving controlled inhalation through the nose and prolonged exhalation into a balloon while maintaining trunk engagement, performed alongside core exercises for eight weeks.
  Arms: Core Stability Training With Balloon Breathing

SUMMARY:
Football players require good core strength and balance to perform well and reduce the risk of injury. The muscles of the trunk and diaphragm play an important role in maintaining stability, posture, and movement control during sports activities.

This randomized controlled trial aims to evaluate the effects of core stability training combined with balloon breathing exercises on dynamic balance, hop performance, and core endurance in professional football players. Balloon breathing exercises are designed to improve diaphragmatic breathing and trunk muscle activation.

Eligible football players will be randomly assigned to one of two groups: one group will receive core stability training combined with balloon breathing exercises along with regular football training, while the other group will receive core stability training with regular football training only. The intervention will be performed three times per week for eight weeks under the supervision of a physiotherapist.

Outcome measures, including dynamic balance, hop performances, core endurance, and maximum voluntary ventilation (MVV), will be assessed at baseline, during the intervention, at the end of the program, and at a three-month follow-up. The findings of this study may help improve training strategies aimed at enhancing performance and reducing injury risk in football players.

ELIGIBILITY:
Inclusion Criteria:

* Male professional football players aged 18 to 35 years
* Currently playing at club level
* Free from musculoskeletal injury for at least 6 months prior to enrollment
* Willing to participate and provide written informed consent
* Able to participate in regular football training and exercise programs

Exclusion Criteria:

* Current musculoskeletal injury or pain affecting training or performance
* History of lower limb or spinal surgery within the past year
* Any neurological, cardiovascular, or respiratory condition that limits physical activity
* Participation in any structured core stability or breathing training program within the past 3 months
* Female players

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Dynamic Balance (Y-Balance Test) | Baseline, 4 weeks, and 8 weeks post-intervention
  Dynamic balance will be assessed using the Y-Balance Test. Reach distances in the anterior, posteromedial, and posterolateral directions will be measured and normalized to leg length.

SECONDARY OUTCOMES:
Core Muscle Endurance | Baseline and 8 weeks
  Core endurance will be assessed using McGill's trunk endurance tests, including trunk flexor hold, trunk extensor hold, and side bridge hold tests. The duration (in seconds) each position is maintained will be recorded.
Lower Limb Hop Performance | Baseline and 8 weeks
  Hop performance will be evaluated using single-leg hop, triple hop, and crossover hop tests. The distance hopped will be measured in centimeters.
Vertical Jump Height | Baseline and 8 weeks
  Vertical jump height will be measured using a validated smartphone application (My Jump 2). The average of the best two out of three trials will be recorded.
maximum voluntary ventilation (MVV) | Baseline and 8 weeks
  Inspiratory muscle strength will be assessed using a portable respiratory pressure meter. The highest value from three maximal inspiratory efforts will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulf medical University, Ajman, Al Jurf, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The effect of core stability training on ball-kicking velocity, sprint speed, and agility in adolescent male football players — https://pubmed.ncbi.nlm.nih.gov/38905315/
- See also: Core stability training for injury prevention — https://pubmed.ncbi.nlm.nih.gov/24427426/
- See also: Effects of neuromuscular training on athletes physical fitness in sports: A systematic review — https://pubmed.ncbi.nlm.nih.gov/36213248/
- See also: Effects of McGill stabilization exercises and conventional physiotherapy on pain, functional disability and active back range of motion in patients with chronic non-specific low back pain — https://pubmed.ncbi.nlm.nih.gov/29706690/
- See also: Revisiting the continuum model of tendon pathology: what is its merit in clinical practice and research? — https://pubmed.ncbi.nlm.nih.gov/27127294/
- See also: Management of patellar tendinopathy: a systematic review and network meta-analysis of randomised studies — https://pubmed.ncbi.nlm.nih.gov/34900334/
- See also: Treatment of patellar tendinopathy--a systematic review of randomized controlled trials — https://pubmed.ncbi.nlm.nih.gov/22186923/